CLINICAL TRIAL: NCT07308379
Title: A Prospective, Observational, Multi-Center, Real-World Study of Toripalimab Injection in First-Line Treatment of Extensive-Stage Small Cell Lung Cancer
Brief Title: Real-World Study of Toripalimab in Extensive-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Other Study IDs: ES-SCLC-01
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: SCLC, Extensive Stage; Toripalimab
Keywords: Extensive stage SCLC; Toripalimab; Real-World Study
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Toripalimab group
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — A humanized IgG4 monoclonal antibody against programmed cell death protein 1 (PD-1). The recommended dosage is 240 mg administered intravenously on Day 1 of each 3-week cycle (q3w). Treatment continues until disease progression, unacceptable toxicity, death, withdrawal of consent, or investigator decision. It is used in combination with chemotherapy (etoposide and platinum-based drugs) as per routine clinical practice.

SUMMARY:
This is a prospective, observational, multi-center, real-world study evaluating the effectiveness and safety of Toripalimab (a PD-1 inhibitor) as first-line treatment for patients with extensive-stage small cell lung cancer (ES-SCLC). The primary objective is to assess real-world progression-free survival (rwPFS). Secondary objectives include evaluating real-world objective response rate (rwORR), disease control rate (rwDCR), overall survival (rwOS), and safety. Approximately 1200 patients from multiple centers in China will be enrolled and followed according to routine clinical practice. Data will be collected from medical records and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate and sign the informed consent form.
* Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC);
* Scheduled to receive Toripalimab as first-line treatment;
* Availability of traceable medical history records during the treatment period.

Exclusion Criteria:

* Pregnant or lactating women;
* Known allergic to recombinant humanized anti-PD-1 monoclonal antibody drugs or their components；
* Any other condition deemed by the investigator as unsuitable for inclusion in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are collected in several hospitals in shanghai, China, diagnosed with extensive-stage small cell lung cancer (ES-SCLC)
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Real-world Progression-Free Survival (rwPFS) | 2 years
  The time from the initiation of the first dose until the first documented occurrence of disease progression or death from any cause, whichever occurs first. Patients who do not experience any event during follow-up or study treatment will be censored at the time of their last tumor assessment. Patients who do not have any post-baseline assessment will be censored on the date of enrollment/initiation of medication.

SECONDARY OUTCOMES:
Real-world Overall Survival (rwOS) | 2 years
  The time from the initiation of the first dose until the documented event of death from any cause. Patients who do not experience the event will be censored at the date of their last known survival. Patients who do not provide any follow-up information will be censored on the date of enrollment/initiation of medication.
Real-world Objective Response Rate (rwORR) | 2 years
  The proportion of patients who achieve a Complete Response (CR) or Partial Response (PR); response is determined by the investigator based on clinician-cited evidence or records without a source of evidence.
Real-world Disease Control Rate (rwDCR) | 2 years
  The proportion of patients who achieve a Complete Response (CR) or Partial Response (PR) or Stable Disease (SD); response is determined by the investigator based on clinician-cited evidence or records without a source of evidence.
Treatment-related adverse event (TRAE) | 2 years
  Including immune-related adverse events (irAEs), particularly Grade ≥3 TRAEs. Monitoring for adverse events will be conducted during the treatment period and until 30 days after the last dose, or until the event resolves or stabilizes.